CLINICAL TRIAL: NCT07021690
Title: Timing Insulin for Meals Using AID Systems
Brief Title: The Steno Opti-Bolus-Timing Studies
Acronym: OBT Studies
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Steno Diabetes Center Copenhagen (Other)
Responsible Party: Principal Investigator, Kirsten Nørgaard, MD, DMSc, Steno Diabetes Center Copenhagen
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Copenhagen University Hospital
Record Dates: First submitted 2025-05-23; First posted 2025-06-15 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Type 1 Diabetes (T1D)
Keywords: AID system; bolus timing; Glycemic index
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: the study contains two sub-studies: breakfast and lunch
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Start high-GI (Active Comparator): T=0: having already rested for 30 min, the participant continues to rest T=15: meal bolus for high GI meal, meal starts T=30: meal ends
  Interventions: Other: High glyceamic index meal
- Pre high-GI (Experimental): T=0: meal bolus for high GI meal T=15: meal starts T=30: meal ends
  Interventions: Other: High glyceamic index meal
- Post high-GI (Experimental): T=0: having already rested for 30 min, the participant continues to rest T=15: meal starts T=30: meal ends T=45: meal bolus for high GI meal
  Interventions: Other: High glyceamic index meal
- Pre low-GI (Experimental): T=0: meal bolus for low GI meal T=15: meal starts T=30: meal ends
  Interventions: Other: Low glyceamic index meal
- Start low-GI (Experimental): T=0: having already rested for 30 min, the participant continues to rest T=15: meal bolus for low GI meal, meal starts T=30: meal ends
  Interventions: Other: Low glyceamic index meal
- Post low-GI (Experimental): T=0: having already rested for 30 min, the participant continues to rest T=15: meal starts T=30: meal ends T=45: meal bolus for low GI meal
  Interventions: Other: Low glyceamic index meal

INTERVENTIONS:
Other: High glyceamic index meal — Meal sizes are standardized regarding the amount of carbohydrate, always 50 g. The composition of these meals focuses on selecting carbohydrates with high glycemic index.
  Arms: Post high-GI; Pre high-GI; Start high-GI
Other: Low glyceamic index meal — Meal sizes are standardized regarding the amount of carbohydrate, always 50 g. The composition of these meals focuses on selecting carbohydrates with low glycemic index.
  Arms: Post low-GI; Pre low-GI; Start low-GI

SUMMARY:
The project investigates the significance of the timing of insulin dosing for breakfast and lunch with an automated insulin pump and whether it matters if the meal primarily contains high or low glycemic index carbohydrates.

We hypothesise that a bolus given 15 minutes before the meal will result in the best blood glucose levels after the meal, regardless of the type of carbohydrates.

Participants will attend 6 experimental days over a maximum of 3 months, where they will be served either breakfast or lunch at the research site, depending on sub-study (breakfast or Lunch sub-study). Three different bolus timings will be tested, with either rapidly absorbed carbohydrates or slowly absorbed carbohydrates, in a randomized order for each participant. Participants will take insulin for the meal using the bolus calculator in the pump, either 15 minutes before, at the start of the meal, or 30 minutes after the meal. The development in sensor glucose will then be monitored for up to 4 hours after the meal.

ELIGIBILITY:
Inclusion criteria:

Type 1 diabetes ≥ 3 years Age 18-70 years User of the MiniMed 780G for at least 3 months Use of Novorapid insulin in the pump (for a minimum of two weeks) TIR > 70% for minimum of 14 days Use carbohydrate counting and bolus calculation Uploads insulin pump and CGM data to the Carelink Personal database Pump settings: carbohydrate ratio (300-500 rule), active insulin time of ≤ 3 hours and smartguard target glucose of 5.5 or 6.1 mmol/L

Exclusion criteria:

Use of anti-diabetic medicine (other than insulin), corticosteroids or other drugs affecting glucose metabolism during the study period or within 4 weeks prior to study start Diagnosed with gastroparesis Females who are pregnant, breast-feeding Food allergies related to standardized meals Alcohol or drug abuse Inability to understand the individual information and to give informed consent.

Current participation in another clinical trial that, in the judgment of the principal investigator, will compromise the study results

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-06-30 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Change in SG between three meal bolus delivery times for meals with two levels of glycemic index | From -15 min before the meal to 270 min after meal intake
  The primary objective is to compare the change in SG (from -15 min before the meal to the highest SG level measured during 0-270 min after start of meal intake) between three meal bolus delivery times for meals with two levels of glycemic index (GI) (high-GI and low-GI meals, respectively).

SECONDARY OUTCOMES:
Area under the post-meal CGM-curve | From -15 min before the meal to 270 min after meal intake
Difference in amount of insulin given for autocorrections during the post-meal period between the three bolus methods for each type of meal. | From -15 min before the meal to 270 min after meal intake
Distribution of Time Below Range (TBR) | From -15 min before the meal to 270 min after meal intake
  Distribution of TBR in the observation period of 4 hours and 45 minutes around the meal between the three bolus methods for each GI meal.
Difference in the number of Time Below Range events (with SG< 3.9 mmol/l) | From -15 min before the meal to 270 min after meal intake
  Difference in the number of Time Below Range (TBR) events (with SG< 3.9 mmol/l) in the observation period of 4 hours and 45 minutes around the meal between the three bolus methods for each GI meal.
Distribution of Time In target Range (TIR) | From -15 min before the meal to 270 min after meal intake
  Distribution of Time In target Range (TIR) in the 4 hours and 45 minutes observation period around the meal between the three bolus methods for each GI meal.
Distribution of Time In Tight target Range (TITR) | From -15 min before the meal to 270 min after meal intake
  Distribution of Time In Tight target Range (TITR), in the 4 hours and 45 minutes observation period around the meal between the three bolus methods for each GI meal.
Distribution of Time Above Range (TAR) | From -15 min before the meal to 270 min after meal intake
  Distribution of Time Above Range (TAR), in the 4 hours and 45 minutes observation period around the meal between the three bolus methods for each GI meal.
Number of hypoglycemia events (PG< 3.9 mmol/L ) | From -15 min before the meal to 270 min after meal intake

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten Nørgaard, Professor, Principal Investigator — Steno Diabetes Center Copenhagen Clinical Translational Research, Diabetes Technology
Locations (1):
- Steno Diabetes Center Copenhagen Clinical Translational Research, Diabetes Technology, Herlev, Denmark

IPD SHARING:
Plan to Share IPD: No